CLINICAL TRIAL: NCT02208102
Title: Association of Cardiac Biomarkers With AF Ablation
Brief Title: Role of Cardiac Biomarkers in Prediction of Outcome in Atrial Fibrillation Patients Undergoing Catheter Ablation
Acronym: IMPACTII
Status: Completed | Type: Observational
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: TCAI_IMPACT II
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation, catheter ablation, blood-biomarkers
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma from whole blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Radio-frequency catheter ablation
  Other Names: RFCA

SUMMARY:
The purpose of this study is to assess if pre-ablation levels of inflammatory biomarkers serve as independent predictors of procedure outcome To evaluate the inflammatory activation following catheter ablation by measuring serum-biomarker levels 24-hours after the procedure and examine the predictive role in procedure success To study the association of certain biomarkers with specific types of AF (paroxysmal or persistent or long standing persistent)

DETAILED DESCRIPTION:
Specific Aim: The purpose of this prospective study is to evaluate the role of inflammatory biomarkers in predicting procedure-outcome in AF patients undergoing catheter ablation.

Background: AF is the most common arrhythmia in clinical practice, affecting > 2.3 million people in US. It increases dramatically with age and is seen in as many as 9% of individuals by the age of 80 (1). A major cause of stroke, AF is also associated with a 2-fold increase in mortality (1).

Symptomatic AF has been demonstrated to be consistently associated with elevated inflammatory activity in the atrial tissue as evidenced by the facts that AF occurs in 40% of patients following cardiac bypass surgery and 50% of patients undergoing valvular surgery (2). Recent studies have also demonstrated that elevated CRP level can increase the risk of AF up to 31% (2). Oxidative damage experienced during AF leads to myocardial necrosis which in turn induces low-grade inflammation resulting in eventual fibrosis of the atrial myocardium. Thus, inflammation can be responsible for adverse structural and electrical remodeling of the cardiac tissue which can further perpetuate the existence, maintenance, and recurrence of this arrhythmia.

Radiofrequency catheter ablation (RFCA) has evolved as a promising curative therapy for drug-refractory AF. However, the recurrence of AF after RFCA is a common clinical problem, occurring in 25-50% of patients in the follow-up period (3) and some patients undergo multiple ablation procedures before being cured of the arrhythmia. Published retrospective studies have demonstrated that systemic inflammation generated during AF ablation is associated with fewer early arrhythmia recurrences (4). Therefore, measurement of inflammatory markers within 24 hours of RFCA could be helpful in further exploration of any association between the degree of inflammatory activation and procedure outcome.

Myriad Rules-Based Medicine, Inc (Myriad RBM) in Austin, TX 78759 has developed biomarker panels that have been validated to detect early signs of inflammation. Myriad RBM will process the blood samples on a preliminary panel of 77 biomarkers, identified to be possible predictors of procedural outcome in RFCA in AF patients.

Study design:

This study will assess a panel of 77 biomarkers in human serum samples that have been identified by the pilot study results as the potential predictors of procedural outcome in catheter ablation for AF. The study population will consist of 150 volunteering patients with AF undergoing RFCA. Blood samples will be collected at two time points from each patient; one at baseline and the other in the morning after the procedure.

Study Procedure:

For each patient, one 8.5 ml tube of whole blood will be collected via venipuncture before and the morning after the ablation procedure.

Ablation Procedure:

Standard radiofrequency catheter ablation procedure will occur in accordance with the physician's discretion.

Blood sample collection:

The whole blood sample will be collected in a Serum Separator Tube (SST) using BD venipuncture procedure, and labeled with an anonymous patient identifier. Only clinical research staff will be able to identify study participants.

Following collection, the samples will be centrifuged for 15 minutes at 900Xg at room temperature, within two hours of collection. Plasma, located as a clear straw-color fluid at the top of the specimen, would be transferred to another sterile tube and stored at -200 C. Samples will be picked up weekly by the RBM team to be stored at -800 C until the end of the study, when all samples will be simultaneously analyzed.

Limited information will also be recorded such as age, gender, height, weight, caffeine intake and information about medications, smoking history, family history of atrial fibrillation (if known), and information about the outcome of the procedure. Researchers at RBM will be blinded to the patient history and demographic data.

After this study is complete the researchers at RBM will store any leftover blood. The researchers may use the leftover samples in future unspecified research studies, which may or may not be related to the AF procedure. Even if the blood sample is used for other studies, the researchers will not have a way to identify the patient.

Follow-Up:

At the 6 and 12 month time points, information will be collected from the medical record regarding recurrence of AF.

Risk Analysis:

Minor risks associated with a venous blood draw may include fainting or bruising, pain or discomfort and a 1/1000 risk of infection at the site where blood is drawn.

ELIGIBILITY:
Inclusion Criteria:

Age: 50-70 years

* Patients undergoing catheter ablation of atrial fibrillation
* Able and willing to give written consent

Exclusion Criteria:

* Reversible causes of AF such as pericarditis and hyperthyroidism

  * Associated chronic inflammatory diseases such as chronic gingivitis or peri-odontitis, rheumatoid Arthritis, IBD including Ulcerative Colitis and Crohn's disease, Lupus, Ankylosing Spondylitis, COPD, psoriasis, vasculitis
  * Any other co-morbid conditions except Diabetes and hypertension
  * Patients taking long-term anti-inflammatory, steroid medication, or immune suppression medication.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing catheter ablation for atrial fibrillation
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Arrhythmia recurrence | 1 year
  Patients will be monitored for arrhythmia recurrence for 1 year after the ablation procedure. At the end of the study, biomarker data will be analyzed to see any predictive association with AFib recurrence

SECONDARY OUTCOMES:
Left atrial scar | During ablation procedure
  if atrial scar is detected during the first ablation procedure, we will assess the association of scar with any of the 77 biomarkers, specifically those indicating fibrosis

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Cardiac Arrhythmia Institute, St. david's Medical Center, Austin, Texas, United States